CLINICAL TRIAL: NCT06833112
Title: Efficacy and Safety of Interleukin-17 Inhibitor in Combination With Tumor Necrosis Factor α Inhibitor in the Treatment of Ankylosing Spondylitis
Brief Title: Interleukin-17 (IL-17) Inhibitor in Combination With Tumor Necrosis Factor α (TNFα )Inhibitor for the Treatment of Ankylosing Spondylitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024114K
Record Dates: First submitted 2025-01-22; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; Secukinumab; adalimumab
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — secukinumab; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- treatment group (Experimental): The subjects were treated with adalimumab (HS016) in combination with secukinumab
  Interventions: Drug: Secukinumab; Drug: Adalimumab

INTERVENTIONS:
Drug: Secukinumab — The subjects were treated with secukinumab for 104 weeks. Secukinumab:150mg，q8w，subcutaneous injection.
Drug: Adalimumab — The subjects were treated with adalimumab for 104 weeks. adalimumab: 40mg，q4w，subcutaneous injection.

SUMMARY:
The aim of the study is to investigate the efficacy and safety of adalimumab in combination with secukinumab for the treatment of ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years old;
2. diagnosed with AS according to the 1984 New York Modified Criteria;
3. Poor response after at least 2 NSAIDs (cumulative treatment ≥ 4 weeks), or contraindication or intolerance to NSAIDs therapy;
4. BASDAI score of ≥ 4 and total back pain VAS score of ≥ 4 at baseline;
5. Subjects who need to take NSAIDs (including COX-1 or COX-2 inhibitors) as established treatment for AS, and the NSAIDs should be on a stable dose for at least 2 weeks (inclusive) before screening and the dose is expected to be stable during the study;
6. Voluntary treatment with adalimumab and secukinumab;
7. Appropriate contraceptive measures for women of childbearing age;
8. without other rheumatic diseases.
9. Able to understand study requirements, provide written informed consent, and comply with trial protocol procedures (including required visits)

Exclusion Criteria:

1. With unstable vital signs, coma, mental and cognitive impairment;
2. Patients with severe systemic diseases and other serious chronic diseases;
3. Pregnant or lactating patients;
4. History of malignant tumor in the past 5 years;
5. Positive test for the following infection markers: human immunodeficiency virus (HIV), hepatitis B, hepatitis C, syphilis antibody;
6. Patients with active or recurrent history of infection; With active tuberculosis or have a history of active tuberculosis in the past;
7. Moderate to severe heart failure (New York Heart Association grade 3-4);
8. Allergic to any of the components of adalimumab (HS016) or secukinumab;
9. Subjects who are participating in clinical research of other drugs;
10. In addition to the above, the investigator judged that there are other reasons that are not suitable for participating in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of SpondyloArthritis International Society 40 (ASAS 40) | week 52
  Proportion of subjects achieving ASAS 40 at Week 52. ASAS 40 is a response criterion used to evaluate the effectiveness of treatments in patients with ankylosing spondylitis. It measures the percentage of patients who achieve at least a 40% improvement in disease activity.
  Key Components of ASAS40:
  * Patient Global Assessment:Patient's overall assessment of disease activity
  * Pain: Assessment of spinal pain.
  * Function: Measured by the Bath Ankylosing Spondylitis Functional Index (BASFI).
  * Inflammation: Based on morning stiffness severity and duration.
  Calculation:
  A patient is considered an ASAS40 responder if they achieve at least a 40% improvement or an absolute improvement of ≥2 units (on a 0-10 scale) in at least 3 out of 4 domains, with no worsening in the remaining domain.
ASAS40 | week 104
  1. Proportion of subjects achieving ASAS 40 at Week 104. ASAS 40 is a response criterion used to evaluate the effectiveness of treatments in patients with ankylosing spondylitis. It measures the percentage of patients who achieve at least a 40% improvement in disease activity.
  Key Components of ASAS40:
  * Patient Global Assessment:Patient's overall assessment of disease activity
  * Pain: Assessment of spinal pain.
  * Function: Measured by the Bath Ankylosing Spondylitis Functional Index (BASFI).
  * Inflammation: Based on morning stiffness severity and duration.
  Calculation:
  A patient is considered an ASAS40 responder if they achieve at least a 40% improvement or an absolute improvement of ≥2 units (on a 0-10 scale) in at least 3 out of 4 domains, with no worsening in the remaining domain.
Modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) | week 104
  The mSASSS is a method used to assess spinal damage and function in patients with ankylosing spondylitis.
  The assessment Items includes:
  * Vertebral Scoring: It evaluates the morphology of each vertebra from T1 to L5. Each vertebra is scored from 0 to 3 based on the presence and degree of squaring, erosions, and syndesmophytes. For example, 0 means normal vertebra, and 3 indicates severe structural changes.
  * Intervertebral Disc Scoring: The intervertebral discs between the vertebrae are also assessed. The score ranges from 0 to 2, depending on the presence and extent of disc space narrowing and bridging syndesmophytes.
  Total Score Calculation: The scores of all vertebrae and intervertebral discs are summed up to obtain the mSASSS total score. The higher the score, the more severe the spinal damage.
Spondyloarthritis Research Consortium of Canada (SPARCC) | week 104
  The SPARCC assessment method is a valuable tool in the field of spondyloarthritis research and diagnosis.
  The assessment Items include:
  * Sacroiliac Joint Assessment: It evaluates the sacroiliac joints using magnetic resonance imaging (MRI). The assessment includes aspects such as bone marrow edema, erosion, and fatty infiltration in the sacroiliac joints. Each feature is scored based on its severity and extent.
  * Spinal Assessment: For the spine, SPARCC also uses MRI to assess inflammation. It focuses on detecting signs like vertebral corner inflammation (enthesitis) and discitis. Similar to the sacroiliac joint assessment, specific features are scored according to their characteristics.
  Scoring System: The total SPARCC score is obtained by summing up the scores of different items. Higher scores indicate more severe inflammation and greater disease activity.

SECONDARY OUTCOMES:
Assessment of SpondyloArthritis International Society 20 (ASAS20) | week 12, week 24, week 52
  Proportion of subjects achieving ASAS 40 at week 12, week 24, week 52. ASAS 20 is a response criterion used to evaluate the effectiveness of treatments in patients with ankylosing spondylitis. It measures the percentage of patients who achieve at least a 20% improvement in disease activity.
  Key Components of ASAS20: -Patient Global Assessment:Patient's overall assessment of disease activity -Pain: Assessment of spinal pain. -Function: Measured by the Bath Ankylosing Spondylitis Functional Index (BASFI). -Inflammation: Based on morning stiffness severity and duration.
  Calculation: A patient is considered an ASAS20 responder if they achieve at least a 20% improvement or an absolute improvement of ≥1 units (on a 0-10 scale) in at least 3 out of 4 domains, with no worsening in the remaining domain.
Assessment of SpondyloArthritis International Society 5/6 (ASAS5/6) | week 12, week 24, week 52
  Proportion of subjects achieving ASAS5/6 at week 12, week 24, week 52. A patient is considered an ASAS5/6 responder if they achieve at least a 20% improvement in at least five of the six items mentioned below：
  * Patient's Global Score: The patient's overall pain level is assessed by the Visual Analogue Score (VAS).
  * Patient's nocturnal back pain and overall back pain VAS score: special attention is paid to the condition of nocturnal back pain.
  * BASFI (Bath Ankylosing Spondylitis Functional Index): Evaluates the patient's ability to perform daily activities, such as wearing socks, bending over to pick up objects, etc.
  * Inflammatory response: by the mean score of inflammatory indicators and morning stiffness time in BASDAI (Bath Ankylosing Spondylitis Disease Activity Index).
  * CRP (C-reactive protein): assesses the level of inflammatory markers.
  * Spinal range of motion: By measuring the range of motion of the spine, such as scoliosis.
Assessment in Ankylosing Spondylitis international Society Partial Release (ASAS PR) | week 12, week 24, week 52
  Proportion of subjects achieving ASAS PR at week 12, week 24, week 52 (The absolute score for each of the 4 indicators identified in ASAS 40 ≤ 2 units)
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 | week 12, week 24, week 52
  Proportion of subjects achieving BASDAI 50 at week 12, week 24, week 52. BASDAI50 is defined as a patient who has at least a 50% improvement from baseline in BASDAI score over the course of treatment.
  Assessment Domains (each scale from 0 to 10, the higher the score, the more severe the symptom):
  * Fatigue: Patients are asked to rate their level of fatigue in the past week.
  * Spinal Pain: score the average spinal pain they have experienced in the past week.
  * Joint Pain/Swelling: Patients rate the degree of pain and swelling in their joints in the past week.
  * Localized Tenderness: The pain at the sites where tendons and ligaments attach to bones is evaluated.
  * Morning Stiffness: This is divided into two parts: duration and severity.
  Scoring Calculation:
  The scores of the five aspects above are added together, resulting in a total score ranging from 0 to 50. This total score is then divided by 5 to obtain the final BASDAI score, which ranges from 0 to 10.
BASDAI | week 12, week 24, week 52
  Change from baseline in BASDAI score at week 12, week 24, week 52.
  Assessment Domains (each scale from 0 to 10, the higher the score, the more severe the symptom):
  * Fatigue: Patients are asked to rate their level of fatigue in the past week.
  * Spinal Pain: score the average spinal pain they have experienced in the past week.
  * Joint Pain/Swelling: Patients rate the degree of pain and swelling in their joints in the past week.
  * Localized Tenderness: The pain at the sites where tendons and ligaments attach to bones is evaluated.
  * Morning Stiffness: This is divided into two parts: duration and severity.
  Scoring Calculation:
  The scores of the five aspects above are added together, resulting in a total score ranging from 0 to 50. This total score is then divided by 5 to obtain the final BASDAI score, which ranges from
Bath Ankylosing Spondylitis Functional Index (BASFI) | week 12, week 24, week 52
  Change from baseline in BASFI score. The BASFI assesses a patient's ability to perform 10 daily activities. These include things like bending to pick up an object from the floor, getting in and out of a car, and turning around in bed.
  Scoring Process
  * Each activity is scored on a scale from 0 to 10. A score of 0 means the patient can perform the activity without any difficulty, while a score of 10 indicates that the patient is completely unable to do the activity.
  * After scoring each activity, the scores are added together. The sum ranges from 0 to 100.
  * This sum is then divided by 10 to get the final BASFI score, which ranges from 0 to 10.
  The lower the score, the lower the disease activity.
Visual Analogue Scale (VAS) | week 12, week 24, week 52
  Change from baseline in VAS score. The VAS (Visual Analogue Scale) scoring method is a commonly used tool for quantitative assessment in medicine that allows patients to directly mark their perceived degree of a certain symptom or condition on a straight line. It transforms subjective feelings into objective numerical values for quantification and comparison.
  Scoring Process: a 10-cm straight line is used, with the left end marked as 0 representing no symptom or the best condition, and the right end marked as 10 representing the most severe symptom or the worst condition.
Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) | week 12, week 24, week 52
  The Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) is used to evaluate enthesitis in patients with ankylosing spondylitis.
  Evaluation Sites:The MASES assesses 13 enthesis sites, namely the left and right first costochondral joints, the left and right seventh costochondral joints, the left and right posterior superior iliac spines, the left and right anterior superior iliac spines, the left and right iliac crests, the proximal insertions of the left and right Achilles tendons, and the fifth lumbar spinous process.
  Scoring Criteria:Absence of pain at the enthesis site is scored as 0, and presence of pain is scored as 1. The total score is the sum of the scores of all sites, ranging from 0 to 13.
tender joint count (TJC), swollen joint count(SJC) | week 12, week 24, week 52
  Change from baseline in 44 TJC and 44 TJC
Ankylosing Spondylitis Disease Activity Score based on C-reactive Protein (ASDAS-CRP) | week 12, week 24, week 52
  Change from baseline in ASDAS-CRP. Components of Assessment: 1)Patient Global Assessment : Patients rate their overall disease activity in the past week on a 0 - 100 mm Visual Analogue Scale, with 0 indicating no disease activity and 100 representing the most severe activity.2)Spinal Pain: The patient assesses the pain in the spine in the past week on a 0 - 100 mm VAS, where 0 means no pain and 100 is the most intense pain.3) Inflammatory Back Pain: It is scored based on a binary scale, 0 for no pain.4)C-reactive Protein level.
  Calculation of the Score:
  The ASDAS-CRP score is calculated through a specific formula: ASDAS-CRP = 0.12 × PGA + 0.28 × spinal pain + 0.16 × IBP + 0.10 × ln(CRP + 1). The result of the calculation is the ASDAS-CRP score, which is used to classify the disease activity level. Generally, a score of <1.3 indicates inactive disease, 1.3 - 2.1 indicates low disease activity, 2.1 - 3.5 indicates moderate disease activity, and >3.5 indicates high disease activity.
Ankylosing Spondylitis Disease Activity Score based on Erythrocyte Sedimentation Rate (ASDAS-ESR) | week 12, week 24, week 52
  Change from baseline in ASDAS-ESR. Assessment Elements: 1)Patient Global Assessment: Similar to ASDAS-CRP, patients rate their overall disease activity in the past week on a 0 - 100 mm Visual Analogue Scale (VAS), with 0 meaning no disease activity and 100 being the highest level of activity.2)Spinal Pain: Patients assess their spinal pain in the past week on a 0 - 100 mm VAS, where 0 represents no pain and 100 is the worst pain.3)Inflammatory Back Pain (IBP): It is scored as 0 for no IBP and 1 for having IBP.4)Erythrocyte Sedimentation Rate (ESR): The ESR value in mm/h is used as a key indicator.
  Score Calculation:The formula for calculating ASDAS-ESR is: ASDAS-ESR = 0.12 × PGA + 0.28 × spinal pain + 0.16 × IBP + 0.08 × ln(ESR + 1). The calculated score is used to determine the disease activity level. Typically, a score of <1.3 suggests inactive disease, 1.3 - 2.1 indicates low disease activity, 2.1 - 3.5 represents moderate disease activity, and >3.5 means high disease activity.
Ankylosing Spondylitis Quality of Life (ASQoL) | week 12, week 24, week 52
  Change from baseline in ASQoL. The ASQoL questionnaire consists of 19 questions covering various aspects such as pain, physical function, mental state, and social life. For example, questions about the impact of the disease on daily activities like dressing, walking, and climbing stairs; how the disease affects mood, sleep, and relationships with others.
  Scoring Method: Each question is scored on a 5-point scale, usually from 0 to 4, with 0 indicating no impact on quality of life and 4 indicating a very severe impact. The scores of all questions are summed up. The total score ranges from 0 to 76. A higher score indicates a poorer quality of life.
Adverse event (AE) | week 12, week 24, week 52，week 104
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jiashun Zeng, Medical Doctor, Principal Investigator — The Affiliated Hospital Of Guizhou Medical University
Locations (1):
- The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No